CLINICAL TRIAL: NCT05918692
Title: A Phase 1, Open-label, Dose-escalation, and Dose-expansion Study of BMF-500, an Oral Covalent FLT3 Inhibitor, in Adults With Acute Leukemia
Brief Title: A Phase 1 Study of BMF-500 in Adults With Acute Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biomea Fusion Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVALENT-103
Record Dates: First submitted 2023-05-18; First posted 2023-06-26 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: FLT3; FLT3-ITD; FLT-TKD; AML; FLT3 Wild-Type; MLL-R; NPM1; CYP3A4
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Accelerated Titration Design, Followed by Modified 3+3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: Escalation Phase (Experimental): BMF-500 taken twice daily by participants who are not receiving drugs that inhibit CYP3A4 activity.
  Interventions: Drug: BMF-500
- Arm B: Escalation Phase (Experimental): BMF-500 taken twice daily by participants who are receiving necessary azole antifungals that are Strong CYP3A4 inhibitors.
  Interventions: Drug: BMF-500
- Arm C: Escalation Phase (Experimental): BMF-500 taken twice daily by participants who are receiving necessary azole antifungals that are moderate CYP3A4 inhibitors.
  Interventions: Drug: BMF-500

INTERVENTIONS:
Drug: BMF-500 — Investigational Product

SUMMARY:
A Phase 1 first-in-human dose-escalation and dose-expansion study of BMF-500, an oral FLT3 inhibitor, in adult patients with acute leukemia.

DETAILED DESCRIPTION:
A Phase 1 first-in-human dose-escalation and dose-expansion study of BMF-500, an oral covalent FLT3 inhibitor, in adult patients with acute myeloid leukemia (AML), who may or may not be on Antifungals.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years.
* Individuals with histologically or pathologically confirmed diagnosis of relapsed or refractory AML with documented FLT3 mutation, and/or Individuals with histologically or pathologically confirmed diagnosis of their malignancy with wild-type FLT3 (including those with MLL1-R and NPM1 mutations).
* ECOG performance status of 0-2.
* Adequate liver and renal function
* Adhere to the CYP3A4 inhibitor concomitant therapy use requirements, as follows:
* Arm A: Participants must not have received a moderate or strong CYP3A4 inhibitor for at least 7 days prior to enrollment and are not anticipated to require such agents in the near term (for at least 4 weeks).
* Arm B: Participants must have received a necessary azole antifungal(s) that is a strong CYP3A4 inhibitor (excluding other strong CYP3A4 inhibitor[s]) for at least 7 days prior to enrollment and be able to continue such azole antifungal(s) while on BMF-500 treatment for at least 4 weeks.
* Arm C: Participants must have received necessary azole antifungal(s) that are moderate CYP3A4 inhibitors (excluding other moderate CYP3A4 inhibitors) for at least 7 days prior to enrollment and be able to continue such azole antifungal(s) while on BMF-500 treatment for at least 4 weeks (Cycle 1).

Key Exclusion Criteria:

* Significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension or arrhythmia, history of cerebrovascular accident including transient ischemic attack within 6 months prior to the first dose of the trial intervention.
* WBC count >50,000/µL (uncontrollable with cytoreductive therapy).
* Women who are pregnant or lactating or plan to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of BMF-500 by incidence of Treatment Emergent Adverse Events (TEAEs). | At the end of each 28 Day cycle for a maximum of 32 cycles
  Assessed by the NCI CTCAE version 5.0.
Evaluate the safety and tolerability of BMF-500 by incidence of Serious Adverse Events (SAEs). | At the end of each 28 Day cycle for a maximum of 32 cycles
  Assessed by the NCI CTCAE version 5.0.
Determine the recommended Phase 2 Dose (RP2D) of BMF-500. | At the end of 28 day Dose-Limiting Toxicities (DLT) observation Period
  Safety, as determined by Dose-Limiting Toxicities (clinically significant Adverse Event) within each dose level assessed NCI CTCAE version 5.0.
Determine the recommended Phase 2 Dose (RP2D) of BMF-500. | At the end of 28 day Dose-Limiting Toxicities (DLT) observation Period
  Efficacy within each dose level as determined by composite complete remission (CRc).
Determine the recommended Phase 2 Dose (RP2D) of BMF-500. | At the end of 28 day Dose-Limiting Toxicities (DLT) observation Period
  Pharmacovigilance (PK) at each dose level as determined by the maximum plasma concentration (Cmax).
Determine the recommended Phase 2 Dose (RP2D) of BMF-500. | At the end of 28 day Dose-Limiting Toxicities (DLT) observation Period
  Pharmacovigilance (PK) at each dose level as determined by area under the curve plasma concentration from time 0 to last quantifiable concentration (AUClast).

SECONDARY OUTCOMES:
Determine the pharmacokinetics of BMF-500. | At the end of each cycle (each cycle is 28 days in duration) for 7 cycles
  Maximum plasma concentration (Cmax).
Determine the pharmacokinetics of BMF-500. | At the end of Cycle 1 and 2 (each cycle is 28 days in duration)
  Area under the curve plasma concentration from time 0 to last quantifiable concentration (AUClast).
Evaluate the efficacy of BMF-500 | At the end of each cycle (each cycle is 28 days in duration) for a maximum of 32 cycles
  Composite Complete Remission (CRc).
Assess additional evidence of antitumor activity per investigator assessment as per corresponding response criteria. | At the end of each cycle (each cycle is 28 days in duration) for a maximum of 32 cycles
  Duration of Response (DOR).
Evaluate the efficacy of BMF-500 | At the end of each cycle (each cycle is 28 days in duration) for a maximum of 32 cycles
  Overall Reasons Rate (ORR).
Assess additional evidence of antitumor activity per investigator assessment as per corresponding response criteria. | At the end of each cycle (each cycle is 28 days in duration) for a maximum of 32 cycles
  Relapse free survival (RFS).
Assess additional evidence of antitumor activity per investigator assessment as per corresponding response criteria. | At the end of each cycle (each cycle is 28 days in duration) for a maximum of 32 cycles
  Overall Survival (OS).

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Mayo Clinic, Phoenix, Arizona
  - City of Hope National Medical Center, Duarte, California
  - University of California, San Francisco, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Kentucky - Markey Cancer Center, Lexington, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Texas Oncology-PA USOR, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Gainesville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No